CLINICAL TRIAL: NCT06744400
Title: Optimal Dose of Anti-lymphocyte Globulin in Kidney Transplant Recipients With Low Immunological Risk
Acronym: ODORAT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024/874
Record Dates: First submitted 2024-12-02; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Renal Transplantation
Keywords: kidney transplant; anti-lymphocyte globulin; Grafalon; Immunosuppression

STUDY DESIGN:
Intervention Model Description: The number of patients included at each dose is determined according to Bayesian optimal interval (BOIN) design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 3 : 2 mg/kg/j (Experimental): Group 3 receives treatment in accordance with health recommendations as part of prophylactic treatment for acute rejection after allogeneic solid organ transplantation, at the minimum dose, i.e., 2 to 5 mg/kg/day for 5 to 21 days.
  Interventions: Drug: Grafalon® administered during 5 consecutive days at 2 mg/kg/j
- Group 2 : 1 mg/kg/j (Experimental): Group 2 receive treatment at lower doses than the recommended dose for the same duration (5 days).
  Interventions: Drug: Grafalon® administered during 5 consecutive days at 1 mg/kg/j
- Group 1 : 0,5 mg/kg/j (Experimental): Group 1 receive treatment at lower doses than the recommended dose for the same duration (5 days).
  Interventions: Drug: Grafalon® administered during 5 consecutive days at 0,5 mg/kg/j

INTERVENTIONS:
Drug: Grafalon® administered during 5 consecutive days at 2 mg/kg/j — This de-escalation study was planned to investigate 3 doses level of Grafalon® administered during 5 consecutive days, i.e.:
  Group 3 : 2 mg/kg/j, Group 2 : 1 mg/kg/j, Group 1 : 0,5 mg/kg/j.
  Group 3 receives treatment in accordance with health recommendations as part of prophylactic treatment for acute rejection after allogeneic solid organ transplantation, at the minimum dose, i.e., 2 to 5 mg/kg/day for 5 to 21 days.
  Other Names: Group 3
  Arms: Group 3 : 2 mg/kg/j
Drug: Grafalon® administered during 5 consecutive days at 1 mg/kg/j — This de-escalation study was planned to investigate 3 doses level of Grafalon® administered during 5 consecutive days, i.e.:
  Group 3 : 2 mg/kg/j, Group 2 : 1 mg/kg/j, Group 1 : 0,5 mg/kg/j.
  Group 2 receive treatment at lower doses than the recommended dose for the same duration (5 days). Treatment begins on the day of transplantation immediately before the procedure at induction of sedation.
  Other Names: Group 2
  Arms: Group 2 : 1 mg/kg/j
Drug: Grafalon® administered during 5 consecutive days at 0,5 mg/kg/j — This de-escalation study was planned to investigate 3 doses level of Grafalon® administered during 5 consecutive days, i.e.:
  Group 3 : 2 mg/kg/j, Group 2 : 1 mg/kg/j, Group 1 : 0,5 mg/kg/j.
  Group 1 receive treatment at lower doses than the recommended dose for the same duration (5 days). Treatment begins on the day of transplantation immediately before the procedure at induction of sedation
  Other Names: Group 1
  Arms: Group 1 : 0,5 mg/kg/j

SUMMARY:
Antithymocyte globulins (ATG) are the gold standard of induction therapies and are currently used to prevent or treat acute rejection in solid organ transplantation. They induce rapid depletion of immune cells, particularly T lymphocytes. The time to immune reconstitution after ATG is characterized by significant intra- and inter-individual variability in reconstitution of immune cell subpopulations (T and B cells, NK cells, dendritic cells). This variability explains the prolonged T cell lymphopenia observed in some patients, which is a surrogate immune biomarker associated with an increased risk of death after 2 years of renal transplantation and more infections, cancers and atheromatous events. However, ATG also promotes an increase in the proportion of Treg cells. Although the underlying mechanisms are still debated, data from experimental animal models confirm the tolerogenic properties of ATG. ATGs are associated with improved allograft survival without rejection in patients at high immunological risk and are therefore indicated as first-line therapy in this population. In patients at low immunological risk, anti-CD25 monoclonal antibodies (anti-CD25mAb) are recommended as first-line therapy because ATGs are associated with a higher incidence of infections despite their equivalent efficacy in this population compared to anti-CD25mAb. However, neither the dosages nor the treatment duration of ATGs are clearly defined (recommended Grafalon® dosages range from 5 to 2 mg/kg/day for 5 to 21 days) and ATGs remain widely prescribed to allow early withdrawal of corticosteroids. Determination of optimal non-depleting doses of ATG could be of great interest because, in vitro, ATG is able to induce regulatory polarization of naïve T cells even at non-depleting doses. Thus, the use of such doses in patients with low immunological risk may be of interest in clinical practice with respect to anti-CD25mAb, particularly for their pro-regulatory properties and their low cost. This question must be clearly addressed in a pilot clinical study.

The purpose of this study is to find the optimal non-depleting dose (Maximum Tolerated Dose; MTD) of rabbit anti-human T-lymphocyte immunoglobulin (Grafalon®) to prevent the complications associated with prolonged CD4 T cell lymphopenia in low immunological risk renal transplant recipients. The primary outcome for the de-escalation study is the Dose Limiting Toxicity (DLT) defined by a T cell (CD3+) relative depletion above 30 % compared to baseline (Day 0) at the end of the Grafalon® induction treatment (Day 4).

The patients under study are adult receiving first kidney transplantation without a high immunological risk of rejection (african-American ethnicity, presence of a donor-specific antibody, blood group incompatibility, delayed onset of graft function (i.e donor after cardiac death), cold ischemia time >24 hours, anti-HLA immunization (Flow PRA > or = 20%, presence of donor specific antibody before and/or at time of transplantation and with a positive CDC and FXM with historical and/or transplant day sera), bacterial, viral or mycotic and parasitic infections, history of opportunistic infection that required intensive care hospitalization in the two years preceding the transplant, related donor with two-haplotype HLA matched kidneys, multi-organ transplant, history of cancer, thrombocytopenia < 50 000 platelets/µl, hypersensitivity to the active substance or to the excipients of Grafalon (monosodium phosphate dihydrate, phosphoric acid).

The inclusion period is one year. According to the active file of the center of Besançon, it is planned to include 2 patients per month. The maximum number of patients to include is 18. With a margin of error of 20%, it is possible to include all patients in 1 year. The duration of patient participation in the study is 1 year (one-year follow-up). Consequently, the duration of the study is estimated at 2 years (1 year of inclusion and 1 year of follow-up).

ODORAT is a monocenter, open-label, de-escalation phase1b controlled study. The study will be proposed to patients receiving a first kidney transplant and matching the criteria of inclusion. Recruitment will be achieved only in Besançon's transplant unit. The physician gives information on the study and collect informed consent. Then the treatment is assigned according to the dose determined by the dose de-escalation study. The first dose tested is the dose level at 2 mg/kg/day (level 3). This dose is the reference dose according to the current recommendations. The number of patients included at each dose is determined according to Bayesian optimal interval (BOIN) design.

The administration of treatment begin at time of transplantation according to recommendation.

The study will include 11 visits: D0 (baseline) to D4 (primary end point assessement), D7, D14, M1, M3, M6 and M12, to analyze pharmacokinetics of Grafalon and the immune phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Females must be using highly effective contraceptive measures (see Section V-9), and have a negative pregnancy test prior to the start of dosing if of childbearing potential, or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening :

  * Post-menopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
  * Women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution.
  * Women with documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
  * Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study drug. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing study treatment.
* Patient affiliated to or beneficiary of French social security system
* Signed and dates informed consent
* Patient receiving first kidney transplantation

Exclusion Criteria:

* Current participation in a study of an investigational agent or in the period of exclusion
* Pregnant or breast-feeding subjects,
* Patient under guardianship, curatorship or under the protection of justice
* Subject not able to cooperate properly in the study judged by the investigator.
* Patients with bacterial, viral or mycotic and parasitic infections,History of opportunistic infection that required intensive care hospitalization in the two years preceding the transplant
* Patients with a high immunological risk of rejection:

  * African-American ethnicity
  * Presence of a donor-specific antibody
  * Blood group incompatibility
  * Delayed onset of graft function (i.e donor after cardiac death)
  * Cold ischemia time >24 hours
  * Anti-HLA immunization (Flow PRA > or = 20%, presence of donor specific antibody before and/or at time of transplantation and with a positive CDC and FXM with historical and/or transplant day sera)
* Related donor with two-haplotype HLA matched kidneys
* Multi-organ transplant
* Previous transplant(s)
* History of cancer
* Thrombocytopenia < 50 000 platelets/µl
* Hypersensitivity to the active substance or to the excipients of Grafalon (monosodium phosphate dihydrate, phosphoric acid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
The optimal non-depleting dose (Maximum Tolerated Dose; MTD) of rabbit anti-human T-lymphocyte immunoglobulin (Grafalon®) to prevent the complications associated with prolonged CD4 T cell lymphopenia in low immunological risk renal transplant recipients. | From transplantation to the end of treatment at 4 days
  The Dose Limiting Toxicity (DLT) defined by a T cell (CD3+) relative depletion above 30 % compared to baseline (Day 0) at the end of the Grafalon® induction treatment (Day 4).

SECONDARY OUTCOMES:
The tolerance of Grafalon® in each dose level. | From transplantation to the end of the study at 1 year.
  Toxicities: Incidence and grade for Adverse events (AEs), drug related AEs, drug related AE leading to dose reduction or discontinuation during treatment, Serious Adverse Events (SAE) and Suspected Unexpected Severe Adverse Reaction (SUSAR), according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0.
Clearance of Grafalon® during the treatment period and until month-3 in each dose level. | From transplantation to 3 month after first treatment.
  Pharmacokinetic study (clearance of Grafalon) including for each dose level the calculation of the plasmatic clearance evaluated by the air under curve of serum active Grafalon® concentration at day 0 and day 4 and the trough level of Grafalon® at each visit until month-3.
Describe immune profile and immune restauration in each dose level. | From transplantation to 1 year after.
  The absolute count and proportion of different T and B cell subpopulations, Natural Killer (NK) cells, monocytes and neutrophils at each time point.
Describe time to event clinical endpoints since transplantation at each dose level. | From transplation to 1 year after.
  Time to Transplant failure defined as the time since transplantation to either graft loss or death with a functioning graft. Return to dialysis or retransplantation defined graft loss.
  Overall survival defined as the time since transplantation to death. Time to kidney allograft acute rejection defined as the time since transplantation since to kidney allograft acute rejection.
The rate of patients with infection up to 1 year after transplantation in each dose level. | From transplantation to 1 year after
  The infection up to 1 year after transplantation defined by :
  * the onset of a severe bacterial infection: all bacterial infections leading to patient hospitalization)
  * or an opportunistic infection: all types of infections that occur only in patients with an immune system deficiency and never in healthy patients (i.e. pneumocystis, tuberculosis, cryptococcosis, candidosis, Kaposi sarcoma, herpesviridae infections, B EBV lymphoma, HTLV T leukemia, toxoplasmosis, cryptococosis, polyomavirus viremia or disease…)
The number of infections by patients up to 1 year after transplantation in each dose level | From transplantation to 1 year after
  The infection up to 1 year after transplantation defined by :
  * the onset of a severe bacterial infection: all bacterial infections leading to patient hospitalization)
  * or an opportunistic infection: all types of infections that occur only in patients with an immune system deficiency and never in healthy patients (i.e. pneumocystis, tuberculosis, cryptococcosis, candidosis, Kaposi sarcoma, herpesviridae infections, B EBV lymphoma, HTLV T leukemia, toxoplasmosis, cryptococosis, polyomavirus viremia or disease…).
The rate of patients with an atherosclerotic event up to 1 year after transplantation in each dose level | From transplantation to year after
  The atherosclerotic event up to 1 year after transplantation defined by major adverse cardiovascular events defined by coronary artery disease, cerebrovascular disease, peripheral arterial disease of the lower limbs, aortic pathology.
Renal function at 1 year post transplant in each dose level | From transplantation to 1 year after.
  Renal function at 1 year post transplant evaluated by estimated glomerular filtration rate (eGFR) calculated by the creatinine clearance according to the formula CKD-EPI.

IPD SHARING:
Plan to Share IPD: Undecided